CLINICAL TRIAL: NCT04944888
Title: Phase ⅠStudy of GSL Synthetase Inhibitor in Combination With Immune Checkpoint Inhibitor in Treating Patients With Advanced Relapsed or Refractory Hematological Malignancies and Previously Treated Solid Tumors
Brief Title: GSL Synthetase Inhibitor in Combination With Immune Checkpoint Inhibitor in Previously Treated Blood and Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-065
Record Dates: First submitted 2021-06-23; First posted 2021-06-30 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Solid Tumor; Hematologic Malignancy
Keywords: GSL synthetase inhibitor; Immune checkpoint inhibitor; Solid tumor; Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — eliglustat; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Dose 1 (Experimental): Eliglustat 84mg will be administered once daily in patients who are CYP2D6 ultra-rapid metabolizers (URMs), extensive metabolizers (EMs), intermediate metabolizers (IMs), or poor metabolizers (PMs), in the first 14 days and the following every other week until 24 weeks. For patients who still benefit from the trial, eliglustat 84mg will be daily administered every other week to 96 weeks.
  Immune checkpoint inhibitor (physician decided) will be administered intravenously on day 5 or day 15 every 3 weeks. For patients who still benefit from the trial, immune checkpoint inhibitor will be administered every 3 week to 96 weeks.
  Interventions: Drug: Eliglustat; Drug: Immune checkpoint inhibitor
- Experimental Dose 2 (Experimental): Eliglustat 84mg will be administered twice daily in patients who are CYP2D6 ultra-rapid metabolizers (URMs), extensive metabolizers (EMs), or intermediate metabolizers (IMs), or in the first 14 days and the following every other week until 24 weeks. For patients who still benefit from the trial, eliglustat 84mg will be administered twice daily every other week to 96 weeks.
  Immune checkpoint inhibitor (physician decided) will be administered intravenously on day 5 or day 15 every 3 weeks. For patients who still benefit from the trial, immune checkpoint inhibitor will be administered every 3 week to 96 weeks.
  Interventions: Drug: Eliglustat; Drug: Immune checkpoint inhibitor

INTERVENTIONS:
Drug: Eliglustat — Eliglustat will be given to enrolled patients at dose of 84mg daily (dose 1) , and then at dose of 84mg twice daily (dose 2).
Drug: Immune checkpoint inhibitor — immune checkpoint inhibitor (physician decided).

SUMMARY:
Immune checkpoint blockade has made great but unsatisfied success in treating cancers. One important reason is the hijacked HLA (Human Leukocyte Antigen) antigen presentation. Eliglustat could inhibit glycosphingolipids synthesis and restore HLA-I antigen presentation and transform the immunogenicity of tumor cells. Therefore,GSL synthetase inhibitor eliglustat in combination with immune checkpoint inhibitor may explore a new avenue for therapeutic intervention in cancer.

DETAILED DESCRIPTION:
Immune checkpoint blockade has led to great strides in the management of various cancers, however, durable response could be seen in approximately 20% of treated patients with most solid tumors and hematological malignancies. One important reason is that tumor cells often escape from immune surveillance by downregulating one or multiple molecules critical in HLA antigen presentation. As a consequence, options that could restore HLA antigen presentation may augment immune checkpoint inhibitor-mediated immune responses.

Abnormal expression of glycosphingolipid (GSL) synthetase is a basic and specific characteristic of most tumors and tumor microenvironment, such as Globo H Ceramide, which is overexpressed in multiple epithelial-derived tumors. Several studies also reported that GSL synthetase was overexpressed in chemotherapy-resistant tumors. Eliglustat is an orally GlcCer synthase inhibitor, which is approved for treating Type-1 Gaucher disease. However, one most recent study reveals that it could inhibit glycosphingolipids synthesis and restore HLA antigen presentation, and transforming the immunogenicity of tumor cells. Therefore, GSL synthetase inhibitor eliglustat in combination with immune checkpoint inhibitor may explore a new avenue for therapeutic intervention in cancer.

The primary objective of this study is to assess the safety and feasibility of GSL synthetase inhibitor eliglustat in combination with immune checkpoint inhibitor in patients with relapsed or refractory hematological malignancies and solid tumors. The secondary objectives include assessing antitumor activity, pharmacokinetics and pharmacodynamics. The exploratory objectives are to evaluate the pathological, immunological or clinical predictive biomarkers for efficacy and toxicity, transformation of tumor microenvironment and dynamic changes of immune cells in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 16 to 75 years with estimated life expectancy >3 months.
2. Histopathological confirmed advanced or metastatic systematically pretreated solid tumors and relapsed/refractory hematological malignancies.
3. Have at least one measurable target lesion for solid tumors.
4. Fresh solid tumor samples or formalin-fixed paraffin embedded tumor archival samples within 3 months are necessary; Fresh tumor samples are preferred. Subjects are willing to accept tumor re-biopsy in the process of this study.
5. Previous treatment must be completed for more than 4 weeks prior to the enrollment of this study, and subjects have recovered to <= grade 1 toxicity.
6. Have an Eastern Cooperative Oncology Group performance status (ECOG) of 0 or 2 at the time of enrollment.
7. Have adequate organ function, which should be confirmed within 2 weeks prior to the first dose of study drugs.
8. Previous treatment with anti-PD-1/PD-L1 antibodies or cytotoxic T lymphocyte associated antigen 4 (CTLA-4) inhibitors are allowed.
9. Ability to understand and sign a written informed consent document.
10. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, and up to 90 days after the last dose of the drug.

Exclusion Criteria:

1. Patients are unwilling to comply with the requirements of the protocol.
2. The patient has documented prior esophageal varices or liver infarction or current liver enzymes (alanine transaminase, aspartate aminotransferase) or total bilirubin >3 times the upper limit of normal.
3. The patient is known to have any of the following: cardiac disease (congestive heart failure, recent acute myocardial infarction, bradycardia, heart block, ventricular arrhythmia), long QT syndrome, current treatment with Class IA or Class III antiarrhythmic medicinal products, interstitial lung disease of any grade or severely impaired pulmonary function.
4. Uncontrolled intercurrent illness, including ongoing or active systemic infection or psychiatric illness/social situations and any other illness that would limit compliance with study requirements and jeopardize the safety of the patient.
5. The patients is taking a CYP2D6 inhibitor and/or concomitantly with a strong or moderate CYP3A inhibitor.
6. Active, known or suspected autoimmune diseases.
7. Known brain metastases or active central nervous system (CNS). Subjects with CNS metastases who were treated with radiotherapy for at least 3 months prior to enrollment, have no central nervous symptoms and are off corticosteroids, are eligible for enrollment, but require a brain MRI screening.
8. Patients are being treated with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment.
9. History of severe hypersensitive reactions to other monoclonal antibodies.
10. History of allergy or intolerance to study drug components.
11. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
12. History of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
13. Pregnant or breast-feeding. Women of childbearing potential must have a pregnancy test performed within 7 days before the enrollment, and a negative result must be documented.
14. Previous or concurrent cancer within 3 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
15. Vaccination within 30 days of study enrollment.
16. Active bleeding or known hemorrhagic tendency.
17. Subjects with unhealed surgical wounds for more than 30 days.
18. Being participating any other trials or withdraw within 4 weeks.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects occuring treatment related adverse events | Up to 90 days after the last dose of study drugs.
  Determining the safety profile following the initiation of treatment and grading these toxicities by CTCAE v5.0

SECONDARY OUTCOMES:
The percentage of enrolled patients that respond to the treatment | Up to 120 days after the last dose of study drugs
  Overall response rate is defined as the sum of partial responses and complete responses

OTHER OUTCOMES:
Immunological response (cytokines, lymphocyte phenotype) | Up to 120 days after the last dose of study drugs
  Immunological responses, including the concentration of cytokines in tumor beds and peripheral blood and the changes of lymphocyte phenotype following the treatment, will be assessed by qPCR and flow cytometer.
Biomarkers predictive of response and toxicity | Up to 120 days after the last dose of study drugs
  Biomarkers from tumor cells, lymphocytes and tumor microenvironment will be assessed for their potential in predicting clinical response and toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, PhD, Principal Investigator — Biotherapeutic Department, Chinese PLA General Hospital
Locations (1):
- Department of Biotherapeutic, Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No